CLINICAL TRIAL: NCT02463474
Title: Piloting the Acceptability of a Culturally Tailored Evidence-Based mHealth Intervention for Low-Income Black Women With Breast Cancer
Brief Title: Mobile Health (mHealth) Black Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201401002
Record Dates: First submitted 2015-05-29; First posted 2015-06-04 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2017-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- mHealth Intervention (Experimental): Each week for 10 weeks, participants will receive two text messages on their cell phone. The first text message will contain a link to a culturally tailored, informational video clip about living with breast cancer. The second text message that provides a supportive message about the video content.
  Interventions: Behavioral: mHealth Intervention

INTERVENTIONS:
Behavioral: mHealth Intervention — Ten, short, engaging, entertaining and culturally relevant videos delivered to participants' cell phones provide breast cancer health information.

SUMMARY:
This research study will test whether a series of video clips with breast cancer information improves knowledge of breast cancer, breast cancer treatment and living with breast cancer. Questionnaires will be completed to learn if the videos are helpful and pleasant to watch.

DETAILED DESCRIPTION:
Though Black women have a lower breast cancer rate than White women, Black women have the poorest outcomes of all races and ethnicities. Low cancer knowledge and mistrust of the healthcare system have been shown to lead to poorer outcomes following breast cancer diagnosis. Participants are asked to be in this research study if they are a woman age 21 years or older who identifies as Black/ African American and has been diagnosed with breast cancer within the past 6 months.

First, participants will come to a pre-intervention study appointment and will be asked to complete several questionnaires. The questionnaires will ask about breast cancer knowledge, quality of life, and their relationship with their doctor. Participants will then opt-in to the study by sending a text message to the study.

For the next ten ten weeks, participants will receive a text message with a link to one video clip per week. Each video is 15-20 minutes long and contains information about breast cancer. Participants will also receive one supportive text message per week for ten weeks.

At the end of the ten weeks, participants will be scheduled for a follow-up appointment. Participants will again be asked questions about breast cancer knowledge, quality of life, and their relationship with their doctor. Participants will also be asked what was helpful and not helpful about the videos.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 years or older
* Race/Ethnicity: Black from any cultural background (e.g., African American, Caribbean Islander, Haitian, Black Hispanic, etc.)
* Diagnosed with breast cancer stages 0-III in the past 6 months
* Life Expectancy: ≥12 months
* Income: at or below 200% of the federal poverty line
* Have access to a cellphone
* Able to receive text messages on cell phone
* Able to view video clips on cell phone.

Exclusion Criteria:

* Previous diagnosis of any type of cancer
* Conditions or behaviors likely to affect the conduct of the trial: unwilling or unable to give informed consent; unable to understand spoken English at the 8th grade level; unwilling to travel to University of Florida Health Shands hospital or HealthStreet for baseline and follow-up assessment appointments; inpatient psychiatric treatment for major psychiatric disorder in the past year; substance use disorder in the past year; and other conditions which in the opinion of study staff would adversely affect participation in the trial.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Knowledge | Baseline assessment (Week 1) to post-intervention assessment (Week 10)
  Breast cancer knowledge will be assessed using the Knowledge subscales of the Breast Cancer Surgery Decision Quality Instrument, short version 2 (BCS-DQI, SV2) developed by Massachusetts General Hospital. The knowledge subscale has twelve multiple choice or fill in the blank items about breast cancer, treatment options, recurrence, survival and side effects.

SECONDARY OUTCOMES:
Perceived Involvement in Care Scale | Baseline assessment (Week 1) to post-intervention assessment (Week 10)
  The Perceived Involvement in Care Scale (PICS) is a 13 item self-report scale that assesses patient's perception of doctor and patient behaviors that occur during a medical visit. It assesses the patients' perception of the doctors' facilitation of patient involvement, amount of information exchanged between the patient and doctor, and patient involvement in decision making.
Perceived Stress Scale | Baseline assessment (Week 1) to post-intervention assessment (Week 10)
  The Perceived Stress Scale (PSS) is a 10-item, self-report questionnaire of globally perceived stress. Each item is rated for the past month on a 5-point Likert scale (1 = never to 5 = very often). A higher total score indicates greater stress.
Functional Assessment of Cancer Therapy-Breast (FACT-B) | Baseline assessment (Week 1) to post-intervention assessment (Week 10)
  This questionnaire is a global measure of quality of life. The FACT-B assesses well-being across five broad domains (i.e., physical, spiritual, social/family, emotional, and functional) and one specific domain of breast cancer symptoms. The instructions ask participants to indicate to what degree each statement has been "true" during the past seven days.
Acceptability | Baseline assessment (Week 1) to post-intervention assessment (Week 10)
  This questionnaire queries the participant's ratings of the acceptability of the program. Item content includes: program was a good use of my time, program was helpful, program will be useful in my daily life, program has helped me deal with my breast cancer, likeability of of the interventionist, acceptability of mobile health (mhealth) format, perceived skill of interventionist, ease of participation in intervention, interactions with program staff, ease of trouble shooting difficulties and overall rating

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Ennis Whitehead, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital, Gainesville, Florida, United States